CLINICAL TRIAL: NCT00816842
Title: Plasma Citrulline as Quantitative Biomarker of HIV Associate Villous Atrophy in a Tropical Enteropathy Population
Brief Title: Plasma Citrulline Concentration in Tropical Enteropathy
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Cinzia Papadia, Azienda Ospedaliera Universitaria di Parma
Other Study IDs: EC3184; Prot 84 24/01/06
Record Dates: First submitted 2009-01-02; First posted 2009-01-05 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Malabsorption Syndromes; Granulomatous Enteritis; Enteritis; HIV Enteropathy; Ileal Diseases
Keywords: citrulline; malabsorption; Villous atrophy; enteropathy
MeSH Terms: conditions — Malabsorption Syndromes; Crohn Disease; Enteritis; HIV Enteropathy; Ileal Diseases; Intestinal Diseases

SUMMARY:
Citrulline is an amino acid produced in the intestine and in the liver, but the liver does not contribute significantly to circulating citrulline concentrations. The intestine is thus the only organ that normally releases significant amounts of citrulline into the blood stream. The investigators have designed a study looking at the value of measuring plasma citrulline concentration in patients with tropical enteropathy of mixed HIV status. The focus will be on the ability of the intestine to sustain the individual concerned from a nutritional standpoint. The investigators hypothesise that plasma citrulline concentration is a marker of small bowel absorptive integrity and an appropriate surrogate for HIV related enteropathy.

DETAILED DESCRIPTION:
Preliminary studies reported that plasma citrulline concentrations may be a reliable biochemical marker for intestinal dysfunction and absorptive enterocyte mass. The relationship between citrulline concentration and intestinal function has been supported in other studies including those examining rejection in small bowel allografts. Concentrations of citrulline are dramatically reduced in cases of mucosal damage (e.g. moderate graft rejection or viral enteritis)and strongly correlate (inversely) with severity on biopsy. Plasma citrulline concentration is lower also in patients with villous atrophy (24±13µmol/L)than in healthy subjects (40±10µmol/L)and patients with anorexia nervosa (39±9µmol/L).Experimental studies have been carried out also in assessing the value of citrulline as a marker for severity of small bowel epithelial damage from radiation and viral infections. The plasma citrulline was shown to be a simple, non invasive and sensitive essay to monitor and quantify radiation and/or chemotherapy induced small bowel damage in mice and humans. Otherwise, the literature on citrulline as a potential marker of intestinal and nutritional integrity is young and consistent data for specific conditions as for HIV enteropathy are missing.We hypothesise that plasma citrulline concentration is a marker of small bowel absorptive integrity and an appropriate surrogate for HIV related enteropathy.

ELIGIBILITY:
Inclusion Criteria:

* histologically ascertained Tropical enteropathy
* Mixed HIV status
* Body mass index within normal range

Exclusion Criteria:

* Patients with surgical resection of stomach, duodenum or pancreas; or (UGI) bypass.
* Patients with other important disease, which may interfere with the study (especially diabetes and renal impairment). Alcoholism, drug abuse or any other circumstances, which may compromise the patient's ability to comply with the study requirements.
* Pregnancy
* Patients experiencing diarrhoea within one month since enrolment date
* Use of glucagon-like peptide 2 (GLP2), growth hormone (GH) or glutamine or triglycerides
* Coeliac Disease, Crohn's disease or infectious intestinal disease
* Patients on steroids or FANS
* Oral feeding>1.0-fold the estimated basal metabolic rate as assessed using Harris and Benedict equation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tropical enteropathy with mixed HIV status
Sampling Method: Non-Probability Sample
Dates: Start 1998-10; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
postabsorptive plasma citrulline concentration | within two years since enrolment date

SECONDARY OUTCOMES:
intestinal permeability ratio | within two years since enrolment date

CONTACTS AND LOCATIONS:
Overall Officials: Cinzia Papadia, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Alastair Forbes, BSc MD FRCP ILTM, Study Chair — University College London Hospitals; Antonio Di Sabatino, MD, Study Director — University of Pavia
Locations (1):
- Department of Medicine, University of Zambia School of Medicine, University Teaching Hospital, Lusaka, Lusaka Province, Zambia